CLINICAL TRIAL: NCT02057458
Title: Role of Blood Flow and Vascular Function on Exercise Capacity in Cystic Fibrosis
Brief Title: Blood Flow and Vascular Function in Cystic Fibrosis
Acronym: CF-FLOW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ryan Harris, Assistant Professor, Augusta University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DK100783; R21DK100783 (NIH)
Record Dates: First submitted 2014-02-04; First posted 2014-02-07 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Cystic Fibrosis
Keywords: arterial stiffness; flow-mediated dilation; endothelial function; pulse wave velocity; inflammation; oxidative stress; pulmonary function test; Cystic Fibrosis; Lung Disease; Nitric Oxide; Exercise Capacity; CF; Muscle Function; Sildenafil; Viagra; Revatio
MeSH Terms: conditions — Cystic Fibrosis; Inflammation; Lung Diseases | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acute Study: Sildenafil first, then Placebo (Experimental): In randomized order, on two separate days, endothelial function and exercise capacity will be determined 1 hour following a single dose of sildenafil (50 mg) or placebo.
  Interventions: Drug: Sildenafil (Acute-1 hour); Drug: Placebo
- Acute Study: Placebo first, then Sildenafil (Experimental): In randomized order, on two separate days, endothelial function and exercise capacity will be determined 1 hour following a single dose of sildenafil (50 mg) or placebo.
  Interventions: Drug: Sildenafil (Acute-1 hour); Drug: Placebo
- Sub-Chronic Study Sildenafil (Experimental): Following the acute study, patients will be instructed to take 20 mg of sildenafil, three times a day, for 4 weeks. Endothelial function will be determined within 48 hours following the last dose.
  Interventions: Drug: Sildenafil (Subchronic-4 weeks)

INTERVENTIONS:
Drug: Sildenafil (Acute-1 hour) — Vascular function will be assessed 1 hour following oral ingestion of sildenafil (50 mg)
  Other Names: Viagra; Revatio
  Arms: Acute Study: Placebo first, then Sildenafil; Acute Study: Sildenafil first, then Placebo
Drug: Sildenafil (Subchronic-4 weeks) — Vascular function will be assessed 4 weeks following 20 mg three times per day (TID) of sildenafil for four weeks
  Other Names: Viagra; Revatio
  Arms: Sub-Chronic Study Sildenafil
Drug: Placebo — Sugar pill designed to mimic the sildenafil treatment
  Arms: Acute Study: Placebo first, then Sildenafil; Acute Study: Sildenafil first, then Placebo

SUMMARY:
Cystic fibrosis (CF) has many health consequences. A reduction in the ability to perform exercise in patients with CF is related to greater death rates, steeper decline in lung function, and more frequent lung infections. However, the physiological mechanisms for this reduced exercise capacity are unknown. The investigators laboratory recently published the first evidence of systemic vascular dysfunction in patients with CF. Therefore, it is reasonable to suspect that the blood vessels are involved with exercise intolerance in CF. This study will look at how 1) blood flow and 2) artery function contribute to exercise capacity in CF.

DETAILED DESCRIPTION:
The most disturbing aspect of Cystic Fibrosis (CF) is the associated premature death. Low exercise capacity predicts death in patients with CF and is also associated with a steeper decline in lung function and more lung infections. A critical barrier to improving exercise tolerance in patients with CF is the investigators lack of knowledge regarding the different physiological mechanisms which contribute to their lower exercise capacity. We have compelling data to indicate that the blood vessels may contribute to the low exercise capacity in CF. The impact of this proof of concept investigation will test Phosphodiesterase Type 5 inhibitors (PDE5) inhibitors as a potential therapy in CF and will explore blood flow and endothelial function as potential mechanisms which contribute to exercise intolerance in CF. Improvements in exercise capacity will not only contribute to a better quality of live for patients with CF, it will also increase longevity in these patients.

ELIGIBILITY:
Inclusion Criteria.

* Diagnosis of CF and healthy controls
* Men and women (greater than 18 yrs. old)
* Resting oxygen saturation (room air) greater than 90%
* Forced expiratory volume (FEV1) percent predicted greater than 30%
* Patients with or without CF related diabetes
* Traditional CF-treatment medications
* Ability to perform reliable/reproducible pulmonary function tests (PFT)
* Clinically stable for 2 weeks (no exacerbations or need for antibiotic treatment within 2 weeks of testing or major change in medical status)

Exclusion Criteria.

* Children less than 17 years old
* Body mass less than 20 kg
* A diagnosis of pulmonary arterial hypertension (PAH)
* FEV1 less than 30% of predicted
* Resting oxygen saturation (SpO2) less than 90%
* Self-reported to be a smoker
* Current use of any vaso-active medications
* History of migraine headaches
* Pregnant or nursing at the time of the investigation
* A clinical diagnosis of cardiovascular disease, hypertension, or CF related diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Harris, Ph.D., Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Rodriguez-Miguelez P, Seigler N, Ishii H, Crandall R, McKie KT, Forseen C, Harris RA. Exercise Intolerance in Cystic Fibrosis: Importance of Skeletal Muscle. Med Sci Sports Exerc. 2021 Apr 1;53(4):684-693. doi: 10.1249/MSS.0000000000002521. PMID 33105385
- See also: Laboratory of Integrative Vascular and Exercise Physiology — http://www.livep.net

RESULTS

PARTICIPANT FLOW:
Groups:
- Sub-Chronic Only: participants who were unable to participate in the acute study due to distance from lab but participated in sub-chronic
Period: Recruited for Participation
Arm/Group | Acute Study: Sildenafil First, Then Placebo | Acute Study: Placebo First, Then Sildenafil | Sub-Chronic Only
Started | 8 | 8 | 3
Completed | 8 | 8 | 3
Not Completed | 0 | 0 | 0
Period: Met Inclusion Criteria
Arm/Group | Acute Study: Sildenafil First, Then Placebo | Acute Study: Placebo First, Then Sildenafil | Sub-Chronic Only
Started | 8 | 8 | 3
Completed | 8 | 7 | 3
Not Completed | 0 | 1 | 0
Not completed — Prior history of migraine headaches | 0 | 1 | 0
Period: Acute Study (1 Hour): First Intervention
Arm/Group | Acute Study: Sildenafil First, Then Placebo | Acute Study: Placebo First, Then Sildenafil | Sub-Chronic Only
Started | 8 | 7 | 0
Completed | 6 | 7 | 0
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Period: Acute Study (1 Hour): Second Int.
Arm/Group | Acute Study: Sildenafil First, Then Placebo | Acute Study: Placebo First, Then Sildenafil | Sub-Chronic Only
Started | 6 | 7 | 0
Completed | 6 | 7 | 0
Not Completed | 0 | 0 | 0
Period: Sub-Chronic Study (4 Weeks)
Arm/Group | Acute Study: Sildenafil First, Then Placebo | Acute Study: Placebo First, Then Sildenafil | Sub-Chronic Only
Started | 6 | 7 | 3
Completed | 5 | 7 | 3
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Baseline characteristics reported for the overall study
Arm/Group | Overall Study
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Height [Mean (Standard Deviation); unit: cm] | 160 (13)
Weight [Mean (Standard Deviation); unit: kg] | 54 (17)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 20.4 (4.0)
Body fat [Mean (Standard Deviation); unit: %] | 28.5 (7.9)
O2 saturation [Mean (Standard Deviation); unit: %] | 98 (1)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 108 (11)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 65 (7)

OUTCOME MEASURES:

1. Primary Outcome: Acute Study: Percentage Flow-Mediated Dilation (FMD)
Description: FMD determined one hour after ingestion of 50 mg Sildenafil or placebo
Time Frame: pre-treatment Baseline and 1 hour post-treatment
Measure: Mean (Standard Deviation); unit: percent flow mediated dilation
Groups:
- Acute Study: Sildenafil: FMD % after acute sildenafil treatment
- Acute Study: Placebo: FMD % after acute placebo
Arm/Group | Acute Study: Sildenafil | Acute Study: Placebo
Number analyzed (Participants) | 13 | 13
percent flow mediated dilation
  Pre | 7.8 (4.3) | 7.7 (4.3)
  Post | 7.3 (4.8) | 6.6 (3.7)

2. Primary Outcome: Baseline Diameter
Description: Brachial Artery Diameter during FMD (pre-occlusion or "baseline")
Time Frame: pre-treatment Baseline and following 4 weeks sub-chronic treatment
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Baseline: "Baseline" artery diameter during FMD taken on preliminary visit before having any treatment.
- Sub-chronic Study: Sildenafil: Baseline artery diameter during FMD after sub-chronic (4 weeks) sildenafil treatment
Arm/Group | Baseline | Sub-chronic Study: Sildenafil
Number analyzed (Participants) | 15 | 15
mm | 3.00 (0.59) | 3.06 (0.60)

3. Primary Outcome: Peak Diameter
Description: Peak Brachial Artery Diameter during FMD (post-occlusion)
Time Frame: pre-treatment Baseline and following 4 weeks sub-chronic treatment
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Baseline: Peak artery diameter during FMD taken on preliminary visit before having any treatment.
- Sub-chronic Study: Sildenafil: Peak artery diameter during FMD after sub-chronic (4 weeks) sildenafil treatment
Arm/Group | Baseline | Sub-chronic Study: Sildenafil
Number analyzed (Participants) | 15 | 15
mm | 3.22 (0.60) | 3.30 (0.60)

4. Primary Outcome: Absolute Change in Diameter
Description: Absolute change in brachial artery diameter taken from the FMD assessment
Time Frame: pre-treatment Baseline and following 4 weeks sub-chronic treatment
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Baseline: Absolute change in artery diameter during FMD taken on preliminary visit before having any treatment.
- Sub-chronic Study: Sildenafil: Absolute change in artery diameter during FMD after sub-chronic (4 weeks) sildenafil treatment
Arm/Group | Baseline | Sub-chronic Study: Sildenafil
Number analyzed (Participants) | 15 | 15
mm | 0.21 (0.12) | 0.27 (0.09)

5. Primary Outcome: FEV1 (% Predicted)
Description: Forced Expiratory Volume in the first second expressed as a percent predicted.
Time Frame: pre-treatment Baseline, 1 hour post-treatment, and following 4 weeks sub-chronic treatment
Measure: Mean (Standard Deviation); unit: percent predicted
Groups:
- Baseline: Baseline measures taken on preliminary visit before having any treatment.
- Acute Study: Sildenafil: FEV1 %predicted after acute sildenafil treatment
- Acute Study: Placebo: FEV1 %predicted after acute placebo
- Sub-chronic Study: Sildenafil: FEV1 %predicted after sub-chronic (4 weeks) sildenafil treatment
Arm/Group | Baseline | Acute Study: Sildenafil | Acute Study: Placebo | Sub-chronic Study: Sildenafil
Number analyzed (Participants) | 15 | 13 | 13 | 15
percent predicted | 81 (16) | 75 (12) | 75 (16) | 82 (15)

6. Primary Outcome: VO2 Peak (Absolute)
Description: absolute (L/min) peak oxygen consumption during maximal exercise test
Time Frame: pre-treatment Baseline, 1 hour post-treatment, and following 4 weeks sub-chronic treatment
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Acute Study: Sildenafil: absolute VO2 peak after acute sildenafil treatment
- Acute Study: Placebo: absolute VO2 peak after acute placebo
- Sub-chronic Study: Sildenafil: absolute VO2 peak after sub-chronic (4 weeks) sildenafil treatment
Arm/Group | Baseline | Acute Study: Sildenafil | Acute Study: Placebo | Sub-chronic Study: Sildenafil
Number analyzed (Participants) | 15 | 13 | 13 | 15
L/min | 1.5 (0.4) | 1.7 (0.5) | 1.6 (0.5) | 1.6 (0.5)

7. Primary Outcome: VO2 Peak (Relative)
Description: relative (mL/kg/min) peak oxygen consumption during maximal exercise test
Time Frame: pre-treatment Baseline, 1 hour post-treatment, and following 4 weeks sub-chronic treatment
Measure: Mean (Standard Deviation); unit: mL/kg/min
Groups:
- Acute Study: Sildenafil: relative VO2 peak after acute sildenafil treatment
- Acute Study: Placebo: relative VO2 peak after acute placebo
- Sub-chronic Study: Sildenafil: relative VO2 peak after sub-chronic (4 weeks) sildenafil treatment
Arm/Group | Baseline | Acute Study: Sildenafil | Acute Study: Placebo | Sub-chronic Study: Sildenafil
Number analyzed (Participants) | 15 | 13 | 13 | 15
mL/kg/min | 28.5 (5.6) | 29.3 (6.1) | 26.8 (6.4) | 29.5 (6.4)

8. Primary Outcome: VO2 Peak (Percent Predicted)
Description: Maximal Oxygen consumption expressed as percent predicted taken from maximal exercise test.
Time Frame: pre-treatment Baseline and 1 hour post-treatment, and 4 weeks sub-chronic treatment
Measure: Mean (Standard Deviation); unit: percent predicted
Groups:
- Acute Study: Sildenafil: VO2 peak %predicted after acute sildenafil treatment
- Acute Study: Placebo: VO2 peak %predicted after acute placebo
- Sub-chronic Study: Sildenafil: VO2 peak %predicted after sub-chronic (4 weeks) sildenafil treatment
Arm/Group | Baseline | Acute Study: Sildenafil | Acute Study: Placebo | Sub-chronic Study: Sildenafil
Number analyzed (Participants) | 15 | 13 | 13 | 15
percent predicted | 72 (12) | 77 (13) | 72 (13) | 75 (12)

9. Primary Outcome: VE Peak
Description: peak ventilation (L/min) during maximal exercise test
Time Frame: pre-treatment Baseline, 1 hour post-treatment, and following 4 weeks sub-chronic treatment
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Acute Study: Sildenafil: VE peak after acute sildenafil treatment
- Acute Study: Placebo: VE peak after acute placebo
- Sub-chronic Study: Sildenafil: VE peak after sub-chronic (4 weeks) sildenafil treatment
Arm/Group | Baseline | Acute Study: Sildenafil | Acute Study: Placebo | Sub-chronic Study: Sildenafil
Number analyzed (Participants) | 15 | 13 | 13 | 15
L/min | 65 (19) | 81 (23) | 77 (24) | 72 (21)

10. Primary Outcome: RER Peak
Description: peak respiratory exchange ratio during maximal exercise test
Time Frame: pre-treatment Baseline, 1 hour post-treatment, and following 4 weeks sub-chronic treatment
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Acute Study: Sildenafil: RER peak after acute sildenafil treatment
- Acute Study: Placebo: RER peak after acute placebo
- Sub-chronic Study: Sildenafil: RER peak after sub-chronic (4 weeks) sildenafil treatment
Arm/Group | Baseline | Acute Study: Sildenafil | Acute Study: Placebo | Sub-chronic Study: Sildenafil
Number analyzed (Participants) | 15 | 13 | 13 | 15
ratio | 1.31 (0.15) | 1.17 (0.12) | 1.22 (0.13) | 1.18 (0.14)

ADVERSE EVENTS:
Time Frame: 2 years, 4 months
Groups:
- Overall Study: Overall Study
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT02057458/Prot_SAP_000.pdf